CLINICAL TRIAL: NCT03531528
Title: A Single-arm Trial to Evaluate the Efficacy of an Aggressive Weight Loss Program With a Ketogenic Induction Phase for the Treatment of Chronic Plaque Psoriasis
Brief Title: Aggressive Weight Loss Program in Chronic Plaque Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Giuseppe Moscati Hospital (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Castaldo, Principal Investigator, San Giuseppe Moscati Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CECN/134
Record Dates: First submitted 2018-04-04; First posted 2018-05-21 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): A 4-week protein-sparing, very low-calorie, ketogenic diet and a subsequent 6-week hypocaloric, low glycemic index, Mediterranean-like diet
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — A 4-week protein-sparing, very low-calorie, ketogenic diet and a subsequent 6-week hypocaloric, low glycemic index, Mediterranean-like diet

SUMMARY:
Chronic plaque psoriasis is frequently associated with obesity and previous studies have shown that a calorie-controlled diet inducing body weight loss improves symptoms and increases the response to pharmacologic treatment. Besides, clinical improvement has been directly correlated with the amount of weight loss. Short-term very low-calorie ketogenic diets are responsible for substantial weight loss and attenuate systemic inflammation to a higher extent than moderately hypocaloric diets. This intervention has been recently demonstrated to restore, after only 4 week, the response to biological therapy in a patient suffering from relapsing moderate-to-severe plaque psoriasis and obesity-related metabolic syndrome. We investigated the efficacy of an aggressive weight loss program with a ketogenic induction phase in a single-arm trial that could provide the rationale for a large randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Stable chronic plaque psoriasis
* Overweight/obese (body mass index >25 kg/m2)

Exclusion Criteria:

* pregnancy and/or lactation
* insulin-dependent diabetes mellitus
* a psychiatric disorder
* current or previous (<1 year since last chemo- or radiotherapy) neoplastic disease
* established vascular disease
* recent (6 months), history of diet-induced or unintentional weight loss
* moderate-to-severe heart failure
* arrhythmia or conduction disorder
* renal failure (creatinine >1.5 mg/dL)
* liver failure (Child-Pugh ≥ A)
* any type of gastrointestinal disease
* moderate-severe hypoalbuminemia (<3.0 g/dL)
* altered serum electrolytes
* refusal to give written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Reduction in Psoriasis Area and Severity Index | 10 weeks
  Change in score (on continuous scale) at the end of study

SECONDARY OUTCOMES:
Reduction in Psoriasis Area and Severity Index | 4 weeks
  Change in score (on continuous scale) at the end of ketogenic diet-phase
Reduction in Psoriasis Area and Severity Index >=75% | 10 weeks
  Proportion of patients with change in score >=75% at the end of study
Reduction in Psoriasis Area and Severity Index >=75% | 4 weeks
  Proportion of patients with change in score >=75% at the end of ketogenic diet-phase
Reduction in Psoriasis Area and Severity Index >=50% | 10 weeks
  Proportion of patients with change in score >=50% at the end of study
Reduction in Psoriasis Area and Severity Index >=50% | 4 weeks
  Proportion of patients with change in score >=50% at the end of ketogenic diet-phase
Reduction in body surface area | 10 weeks
  Change in body surface area (on continuous scale) involved at the end of study
Reduction in body surface area | 4 weeks
  Change in body surface area (on continuous scale) involved at the end of ketogenic diet-phase
Reduction in Dermatology Life Quality Index (DLQI) | 10 weeks
  Change in DLQI (on continuous scale) at the end of study
Reduction in Dermatology Life Quality Index (DLQI) | 4 weeks
  Change in DLQI (on continuous scale) at the end of ketogenic diet-phase
Reduction in itch severity | 10 weeks
  Change in itch severity (on continuous visual analogue scale) at the end of study
Reduction in itch severity | 4 weeks
  Change in itch severity (on continuous visual analogue scale) at the end of ketogenic diet-phase
Reduction in body weight | 10 weeks
  Change in body weight (on continuous scale) at the end of study
Reduction in body weight | 4 weeks
  Change in body weight (on continuous scale) at the end of ketogenic diet-phase
Reduction in Visceral fat | 10 weeks
  Change in aorto-mesenteric fat thickness (on continuous scale) at the end of study
Reduction in Visceral fat | 4 weeks
  Change in aorto-mesenteric fat thickness (on continuous scale) at the end of ketogenic diet-phase

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Castaldo, MD, Principal Investigator — A.O.R.N. "San Giuseppe Moscati", Avellino, Italy
Locations (1):
- A.O.R.N. "San Giuseppe Moscati", Avellino, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Castaldo G, Galdo G, Rotondi Aufiero F, Cereda E. Very low-calorie ketogenic diet may allow restoring response to systemic therapy in relapsing plaque psoriasis. Obes Res Clin Pract. 2016 May-Jun;10(3):348-52. doi: 10.1016/j.orcp.2015.10.008. Epub 2015 Nov 11. PMID 26559897
- [Background] Castaldo G, Monaco L, Castaldo L, Galdo G, Cereda E. An observational study of sequential protein-sparing, very low-calorie ketogenic diet (Oloproteic diet) and hypocaloric Mediterranean-like diet for the treatment of obesity. Int J Food Sci Nutr. 2016 Sep;67(6):696-706. doi: 10.1080/09637486.2016.1186157. Epub 2016 May 18. PMID 27193396
- [Background] Castaldo G, Palmieri V, Galdo G, Castaldo L, Molettieri P, Vitale A, Monaco L. Aggressive nutritional strategy in morbid obesity in clinical practice: Safety, feasibility, and effects on metabolic and haemodynamic risk factors. Obes Res Clin Pract. 2016 Mar-Apr;10(2):169-77. doi: 10.1016/j.orcp.2015.05.001. Epub 2015 Jun 1. PMID 26044613
- [Background] Monaco L, Monaco M, Di Tommaso L, Stassano P, Castaldo L, Castaldo G. Aortomesenteric fat thickness with ultrasound predicts metabolic diseases in obese patients. Am J Med Sci. 2014 Jan;347(1):8-13. doi: 10.1097/MAJ.0b013e318288f795. PMID 24366220